CLINICAL TRIAL: NCT04141319
Title: Effects of Pre-emptive Scalp Infiltration With Ketorolac and Ropivacaine for Postoperative Pain Relief After Elective Supratentorial Craniotomy (PAINLESS)
Brief Title: Effects of Pre-emptive Scalp Infiltration With Ketorolac and Ropivacaine for Post-craniotomy Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Pain Management, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY-2018-034-02-6
Record Dates: First submitted 2019-10-20; First posted 2019-10-28 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Pain; Supratentorial Brain Tumor
MeSH Terms: conditions — Pain | interventions — Ketorolac; Ropivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The ketorolac group (Experimental): Patients assigned to the ketorolac group will receive pre-emptive scalp infiltration with 30ml of local infiltration solution containing 60 mg ropivacaine, 6 mg ketorolac and 0.1mg epinephrine.
  Interventions: Drug: Ketorolac; Drug: Ropivacaine; Drug: Epinephrine
- The control group (Active Comparator): In the control group, preoperative peri-incisional scalp infiltration will be performed using 30ml of 60 mg ropivacaine and 0.1mg epinephrine.
  Interventions: Drug: Ropivacaine; Drug: Epinephrine

INTERVENTIONS:
Drug: Ketorolac — 30ml of local infiltration solution containing 60mg ropivacaine
  Arms: The ketorolac group
Drug: Ropivacaine — 30ml of local infiltration solution containing 6mg ketorolac
Drug: Epinephrine — 30ml of local infiltration solution containing 0.1mg epinephrine

SUMMARY:
The PAINLESS study is a single-center, prospective, randomized, open-label, blinded-endpoint (PROBE) controlled clinical study to compare the efficacy and safety of pre-emptive scalp infiltration with ropivacaine plus ketorolac and ropivacaine alone for postoperative pain relief in adults undergoing elective supratentorial craniotomies.

DETAILED DESCRIPTION:
The proposed study will be a single-center, prospective, randomized, open-label, blinded-endpoint clinical trial designed to test the hypothesis that the addition of ketorolac to pre-emptive scalp infiltration analgesia can significantly improve analgesia after craniotomies. One hundred participants will be randomized to the ketorolac group or the control group. Patients in the ketorolac group will receive pre-emptive scalp infiltration with opivacaine,ketorolac and epinephrine while patients in the control group will receive pre-emptive scalp infiltration with ropivacaine and epinephrine.The primary outcome measure will be cumulative doses of patient-controlled analgesia (PCA) butorphanol consumption from 0 to 48 h postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective supratentorial tumour resection;
* Planned general anaesthesia;
* American Society of Anesthesiologists (ASA) physical status I - II;
* Age ranging from 18 to 65 years old;
* Participates required to fix their head in a head clamp intraoperatively;
* Participates with an anticipated awake within 2 hours after surgery.

Exclusion Criteria:

* Allergy/intolerance to study drugs including anesthetic drugs, ketorolac and epinephrine;
* Expected delayed extubation or no plan to extubate;
* History of neurosurgeries;
* Long-term use of analgesics and sedatives (more than 2 weeks)
* Receiving any painkiller within 24 h before the operation;
* Extreme body mass index (BMI) (less than 15 or more than 35);
* Patients with impaired cardiopulmonary;
* Patients with impaired renal function;
* Patients with impaired hepatic function;
* History of chronic headache;
* Patients with cognitive deficit;
* Patients with intellectual disability;
* Patients with uncontrolled epilepsy;
* Patients with psychiatric disorders;
* Difficulties in using PCA device
* Difficulties in understanding the use of numeral rating scale (NRS) ;
* Patients with suspected intracranial hypertension;
* Pregnant or at breastfeeding;
* Infection at the incisional site；
* History of radiation therapy and chemotherapy preoperatively
* With great likelihood of postoperative radiation therapy and chemotherapy based on preoperative imaging.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
cumulative doses of patient-controlled analgesia (PCA) butorphanol consumption from 0 to 48 h postoperatively | 0 to 48 hours postoperatively
  The primary outcome measure will be cumulative doses of PCA butorphanol consumption from 0 to 48 h postoperatively

SECONDARY OUTCOMES:
The time to first request for patient-controlled analgesia butorphanol | Within 48hours postoperatively
  The time to first request for patient-controlled analgesia butorphanol
frequency of pressing patient-controlled analgesia pump | Within 48hours postoperatively
  frequency of patient-controlled analgesia pump
numeral rating scale (NRS) Score | at 2 hours, 4 hours, 8 hours, 24 hours, 48 hours, 72 hours, 1 week, 2 weeks, 1 month, 3 months and 6 months postoperatively
  0 for"no pain" and 10 for "'pain as severe as you can imagine"
Pain control satisfaction score (PCSS) postoperatively | at 24 hours, 48 hours, 72 hours, 1 week, 1 month, 3 months and 6 months
  0 for unsatisfactory and 10 for very satisfactory
Ramsay sedation score (RSS) | at 2 hours, 4 hours, 8 hours, 24 hours and 48 hours and 72 hours postoperatively
  1: Anxious, agitated, restless; Ramsey 2: Cooperative, oriented, tranquil; Ramsey 3: Responsive to commands only If Asleep; Ramsey 4: Brisk response to light glabellar tap or loud auditory stimulus; Ramsey 5: Sluggish response to light glabellar tap or loud auditory stimulus; Ramsey 6: No response to light glabellar tap or loud auditory stimulus.
  Asleep; Ramsey 4: Brisk response to light glabellar tap or loud auditory stimulus; Ramsey 5: Sluggish response to light glabellar tap or loud auditory stimulus; Ramsey 6: No response to light glabellar tap or loud auditory stimulus.
pulse oxygen saturation(SpO2) | 1 minutes before anesthesia induction, 1 minutes after anesthesia induction, 1 minutes after scalp infiltration, at the beginning of skull drilling, mater cutting and skin closure and at 2hours, 4 hours, 8 hours , 24 hours and 48 hours postoperatively
  SpO2
mean arterial blood pressure(MAP) | 1 minutes before anesthesia induction, 1 minutes after anesthesia induction, 1 minutes after scalp infiltration, at the beginning of skull drilling, mater cutting and skin closure and at 2hours, 4 hours, 8 hours , 24 hours and 48 hours postoperatively
  MAP
heart rate(HR) | 1 minutes before anesthesia induction, 1 minutes after anesthesia induction, 1 minutes after scalp infiltration, at the beginning of skull drilling, mater cutting and skin closure and at 2hours, 4 hours, 8 hours , 24 hours and 48 hours postoperatively
  HR
respiratory rate(RR) | 1 minutes before anesthesia induction, 1 minutes after anesthesia induction, 1 minutes after scalp infiltration, at the beginning of skull drilling, mater cutting and skin closure and at 2hours, 4 hours, 8 hours , 24 hours and 48 hours postoperatively
  RR
Length of hospital stay | Length of hospital stay, an arverage of 2 weeks
  Length of hospital stay
Wound healing score | at 3 weeks and 6 weeks after surgery
  Skin Healing 1: fully healed; 2: ≤3 cm in total not healed; 3: >3 cm not healed; 4: areas of necrosis ≤3 cm; 5: areas of necrosis >3 cm Infection 1: none; 2: ≤0.5-cm margin of redness; 3: more redness or superficial pus; 4: deep infection; not applicable Hair Regrowth 1: even regrowth along wound; 2: ≤3 cm not regrowing; 3: >3-6 cm not regrowing; 4: >6 cm not regrowing; not applicable
postoperative nausea and vomiting(PONV) | within 48 hours postoperatively
  0, absent; 1, nausea but not requiring treatment; 2, nausea requiring treatment; and 3, vomiting
The presence of respiratory depression | within 48 hours postoperatively
  respiratory rate <10 breaths per minute or SpO2 was<90 %
The incidence of haematoma, wound infection or gastric ulcers | during hospitalization, within 2 weeks postoperatively
  side effects

CONTACTS AND LOCATIONS:
Overall Officials: Fang Luo, M.D, Principal Investigator — Beijing Tiantan Hospital

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Vacas S, Van de Wiele B. Designing a pain management protocol for craniotomy: A narrative review and consideration of promising practices. Surg Neurol Int. 2017 Dec 6;8:291. doi: 10.4103/sni.sni_301_17. eCollection 2017. PMID 29285407
- [Background] Andersen KV, Nikolajsen L, Haraldsted V, Odgaard A, Soballe K. Local infiltration analgesia for total knee arthroplasty: should ketorolac be added? Br J Anaesth. 2013 Aug;111(2):242-8. doi: 10.1093/bja/aet030. Epub 2013 Mar 20. PMID 23514638
- [Background] Solovyova O, Lewis CG, Abrams JH, Grady-Benson J, Joyce ME, Schutzer SF, Arumugam S, Caminiti S, Sinha SK. Local infiltration analgesia followed by continuous infusion of local anesthetic solution for total hip arthroplasty: a prospective, randomized, double-blind, placebo-controlled study. J Bone Joint Surg Am. 2013 Nov 6;95(21):1935-41. doi: 10.2106/JBJS.L.00477. PMID 24196463
- [Background] Song J, Li L, Yu P, Gao T, Liu K. Preemptive scalp infiltration with 0.5% ropivacaine and 1% lidocaine reduces postoperative pain after craniotomy. Acta Neurochir (Wien). 2015 Jun;157(6):993-8. doi: 10.1007/s00701-015-2394-8. Epub 2015 Apr 7. PMID 25845547